CLINICAL TRIAL: NCT07081230
Title: Comparison Between the Efficacy of Albumin Versus Hyaluronic Acid Scaffold in Combination With Concentrated Growth Factors as an Adjunct to Non-surgical Treatment of Periodontitis (Randomized Controlled Clinical Trial)
Brief Title: Comparison Between the Efficacy of Albumin Versus Hyaluronic Acid Scaffold in Combination With Concentrated Growth Factors as an Adjunct to Non-surgical Treatment of Periodontitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: husain abduljalil alam (Other)
Responsible Party: Sponsor-Investigator, husain abduljalil alam, Principal Investigator,BDS, Oral Medicine, Periodontology, Diagnosis, and Oral Radiology Department,, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A03010250M
Record Dates: First submitted 2025-07-06; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis | interventions — Hyaluronic Acid

STUDY DESIGN:
Intervention Model Description: Patients will be randomly divided into 3 groups with (10) patients each. Group I (Test group 1): patients will receive hyaluronic acid mixed with concentrated growth factors after mechanical debridement.
  Group II (Test group 2): patients will receive Albumin gel mixed with concentrated growth factors after mechanical debridement.
  Group III (Control group): patients will receive mechanical debridement only.
Masking Description: Randomization will be performed before starting the study by computer generated tables to allocate each patient in his group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HYALURONIC ACID MIX WITH CGF (Experimental): patients will receive hyaluronic acid mixed with concentrated growth factors after mechanical debridement
  Interventions: Combination Product: SRP with hyaluronic acid
- ALB PRF (Experimental): patients will receive Albumin gel mixed with concentrated growth factors after mechanical debridement
  Interventions: Combination Product: SRP + Injectable Platelet-Rich Fibrin

INTERVENTIONS:
Combination Product: SRP with hyaluronic acid — patients will receive hyaluronic acid mixed with concentrated growth factors injected into the periodontal pocket after mechanical debridement
  Arms: HYALURONIC ACID MIX WITH CGF
Combination Product: SRP + Injectable Platelet-Rich Fibrin — patients will receive Albumin gel mixed with concentrated growth factors injected into the periodontal pocket after mechanical debridement
  Arms: ALB PRF

SUMMARY:
The primary objective is to clinically evaluate the efficacy of albumin versus hyaluronic acid scaffolds in combination with concentrated growth factors in the non- surgical treatment of stage II/III periodontitis.

The secondary objective is to evaluate the duration and concentration of different growth factors release in the gingival crevicular fluid.

DETAILED DESCRIPTION:
III. Treatment Procedures:

Three weeks prior to treatment all patients will receive phase I periodontal therapy in the form of non-surgical mechanical debridement using ultrasonic and hand instruments, oral hygiene instructions will be demonstrated to all patients.

Group I (Test group 1): will receive mechanical debridement and injection of hyaluronic acid mixed with growth factor concentrates in the periodontal pocket, the growth factor concentrates will be prepared by collecting peripheral blood using 9-10 mL tubes without adding any additives, following blood collection, the blood tubes will be placed in a centrifuge for the 8-min ,two to four milliliters of the initial portion of plasma PPP (platelet-poor plasma) is then collected with a syringe and discarded, leaving the other blood portions, the LPCGF (liquid phase concentrated growth factors) from buffy coat is collected then it will be mixed using a female-female connector with hyaluronic acid and injected into the pocket.

Group II (Test group 2) : will receive mechanical debridement and ALB-PRF will be prepared by collecting peripheral blood using 9-10 mL tubes without adding any additives, following blood collection, the blood tubes will be placed in a centrifuge for the 8-min ,Two to four milliliters of the initial portion of plasma (platelet-poor plasma) is then collected with a syringe and placed into a heating device , while the other blood portions (buffy coat, LPCGF, and red blood cells) are placed in a cooling storage bag. The syringes containing PPP are then inserted into a heating device for human serum albumin denaturation plasma to produce the albumin gel. After 10 minutes at an operating temperature of 75°C, the syringes are then removed and allowed to cool in a cooling storage bag and protected from ambient light. The LPCGF (liquid phase concentrated growth factors) from buffy coat are then collected. Thereafter, the albumin gel and the liquid-CGF are mixed between syringes by passing back and forth (roughly 10×) using a female-female connector to create ALB-PRF which is ready to be injected in the periodontal pocket, ALB-PRF gel will be injected into periodontal pocket by special needle until it is full.

Group III (Control group): will receive mechanical debridement only. All patients will be advised not to eat hard food, they were also advised not to brush the area for 12h or to floss or use interproximal cleaning devices for ten days. During the study period, the patients were instructed to continue regular tooth brushing and interdental cleansing, also instructed not to use any mouth washes for the Duration of the study.

ELIGIBILITY:
ii) Inclusion Criteria:

* Patients aging from 25-45 years
* Patients with stage II /III periodontitis
* Systemically free iii) Exclusion Criteria:
* Any systemic condition that may impact the study (21)
* Poor oral hygiene
* Pregnant and breastfeeding women
* Smoking patients.
* Patients received periodontal treatment in the last 6 months
* Unable to comply with study protocol

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Plaque index (PI) | baseline, 6weeks, 12weeks
  1. Plaque index (PI):The index assigns a score to each tooth based on the amount of plaque present.
  0: No plaque is visible.
  1. A thin film of plaque is present at the gingival margin (gumline) and can be detected with a probe.
  2. Visible plaque along the gingival margin.
  3. Heavy plaque accumulation in the gingival margin and interdental spaces.
Bleeding on probing (BOP) | baseline, 6weeks, 12weeks
  "0" if no bleeding occurred within 10 second, and "1" if there was bleeding within 10 second.
Probing pocket Depth (PPD) | baseline, 6weeks, 12weeks
  will be measured from the gingival margin to the base of the periodontal pocket
Clinical Attachment Level (CAL) | baseline, 6weeks, 12weeks
  will be measured from the cement-enamel junction to the base of the periodontal pocket

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura university Faculty of dentistry, Al Mansurah, Mansoura, Egypt

IPD SHARING:
Plan to Share IPD: Undecided